CLINICAL TRIAL: NCT03908125
Title: A Post- Approval Study to Evaluate the Long-term Safety and Effectiveness of the Eversense® Continuous Glucose Monitoring (CGM) System
Brief Title: Post Approval Study of the Eversense® Continuous Glucose Monitoring
Acronym: PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-0034
Record Dates: First submitted 2019-03-22; First posted 2019-04-09 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Continuous Glucose Monitoring Device (Other): Commercial Continuous Glucose Monitoring Device
  Interventions: Device: Eversense® CGM System

INTERVENTIONS:
Device: Eversense® CGM System — Continuous Glucose monitoring device

SUMMARY:
A Post Approval Study to Evaluate the Long-term Safety and Effectiveness of the Eversense® Continuous Glucose Monitoring (CGM) System over repeat insertion and removal cycles and to demonstrate the long-term safety of the Eversense® CGM System

DETAILED DESCRIPTION:
The purpose of this post-approval study (PAS) is to provide long-term safety and effectiveness of the Eversense CGM System (PMA Application P160048) in the post-market setting. In the premarket setting, the PRECISE II and PRECISION studies demonstrated safety and accuracy of the CGM system in estimating blood glucose levels compared to reference blood glucose analyzer levels to 90 days.

The PROMISE study demonstrated safety and accuracy of the CGM system up to 180 days. This PAS study will provide safety and effectiveness data up to 27 months of repeated use.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has diabetes
2. Subject is greater than 18 years of age

Exclusion Criteria:

1. Subject is critically ill or hospitalized
2. Subject has a known contraindication to dexamethasone or dexamethasone acetate
3. Subjects requiring intravenous mannitol or mannitol irrigation solutions
4. Female subjects who are pregnant, planning on becoming pregnant or nursing
5. Subjects on hybrid closed loop systems or closed loop systems
6. Subjects on other CGM systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Davis, Study Director — Senseonics, Inc.
Locations (17):
- United States (17):
  - Hoag Memorial Hospital Presbyterian/Mary Dick Allen Diabetes Center, Newport Beach, California
  - Denver Endocrinology, Diabetes & Thyroid Center, Englewood, Colorado
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - MODEL Clinical research, Baltimore, Maryland
  - Metro Detroit Endocrinology Center, Dearborn, Michigan
  - Diabetes and Endocrinology Specialists, Inc., Chesterfield, Missouri
  - Albany Medical College, Albany, New York
  - Physicians East, Greenville, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Diabetes & Endocrinology Consultants of Pennsylvania, LLC, Feasterville, Pennsylvania
  - AM Diabetes & Endocrinology, Bartlett, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Clinical Research Solution, LLC, Cypress, Texas
  - Javara, Inc, Houston, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Glucose Monitoring Device: Eversense® CGM system: Continuous Glucose monitoring device that lasts up to 90 days
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring Device
Started | 273 (Inserted with sensor(s))
Completed | 173
Not Completed | 100
Not completed — Withdrawal by Subject | 92
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Population: Subjects enrolled and inserted with the Eversense CGM system
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 259
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 23
  White | 235
  More than one race | 3
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 273
Diabetes Type [Count of Participants; unit: Participants]
  Type 1 | 218
  Type 2 | 55
Years Since Diabetes Diagnosis [Mean (Standard Deviation); unit: years] | 19 (13)
CGM Naive [Count of Participants; unit: Participants] | 71
Diabetes Therapy Regimen [Count of Participants; unit: Participants]
  Non-insulin medications,basal insulin, lifestyle | 10
  Intensive insulin therapy | 263

OUTCOME MEASURES:

1. Primary Outcome: The Long-term Safety of the Eversense CGM Systems Over Repeat Insertion and Removal Cycles in the Post-market Setting.
Description: The primary safety endpoint was the incidence of the composite of infection, secondary procedures to remove the Sensor, or procedure-related adverse events of at least moderate severity, with a performance goal of < 4%.
Time Frame: up to 27 months
Measure: Count of Units; unit: Sensor cycle
Units Other Than Participants: Sensor cycle
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
Number analyzed (Sensor cycle) | 1528
Sensor cycle
  Infection | 5
  Secondary procedure to remove sensor | 24
  Procedure-related adverse event of at least moderate severity | 15

2. Primary Outcome: The Long-term Effectiveness of the Eversense CGM Systems Over Repeat Insertion and Removal Cycles in the Post-market Setting.
Description: The primary effectiveness endpoint was Time in Range, which is defined as glucose values between 70 mg/dL and 180 mg/dL, at 12 months post-first Sensor insertion compared to the first month post-first Sensor insertion.
Time Frame: Baseline and Month 12
Measure: Mean (Standard Deviation); unit: % time in range
Groups:
- Baseline Time in Range: First month post-first sensor insertion
Arm/Group | Baseline Time in Range
Number analyzed (Participants) | 273
% time in range
  Baseline | 62.9 (18.3)
  Month 12 | 62.4 (20.1)

3. Secondary Outcome: The Additional Effectiveness Endpoint of Average Hours of Use Per Day
Time Frame: up to 27 months
Measure: Mean (Standard Deviation); unit: Daily use [hours]
Units Other Than Participants: sensors
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
Number analyzed (sensors) | 1448
Daily use [hours] | 19 (7)

4. Secondary Outcome: The Additional Effectiveness Endpoint of Change in HbA1c Levels at Each 6-month Interval From Baseline
Time Frame: Baseline, Month 6, Month 12, Month 18, and Month 24
Population: Change in HbA1c from Baseline at 6-Month Intervals. Window for 6, 12, and 18-month intervals was ± 30 days. Window for 24-month interval was -30 days to anything greater than 24 months.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
percentage of HbA1c
  Baseline | 0 (0)
  6-month | -0.16 (1.04)
  12-month | -0.14 (0.96)
  18-month | -0.10 (0.96)
  24-month | 0.06 (1.31)

5. Secondary Outcome: Patient Satisfaction With CGM System Use (CGM-SAT Scale)
Description: CGM-Sat is a 44 question, 5-point scale (1 = strongly agree, 5 = strongly disagree); higher scores reflect more satisfaction with CGM.
Time Frame: up to 27 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
score on a scale
  Day 180 | 4.0 (0.5)
  Day 360 | 4.1 (0.5)
  Day 720 | 4.1 (0.5)

6. Secondary Outcome: Patient Reported Diabetes Distress Scale (DDS)
Description: The DDS score over the two-year period. DDS17 is a 17 question, 6-point scale (1 = not a problem, 6 = a very serious problem); lower score depicts less distress with diabetes.
Time Frame: Screening, Day 180, Day 360, and Day 720
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
score on a scale
  Screening | 1.9 (0.8)
  Day 180 | 1.7 (0.7)
  Day 360 | 1.7 (0.7)
  Day 720 | 1.7 (0.7)

7. Secondary Outcome: Success Rate of Insertion Procedures: Overall and by HCP Experience
Description: Success rate was measured for the first 3 insertions for each inserting HCP, the remaining insertions, as well as overall insertions.
Time Frame: up to 27 months
Population: The number analyzed in the first 2 rows are the subsets of the overall insertions based on HCP experience.
Measure: Number; unit: percentage of successful insertion
Units Other Than Participants: sensor insertions
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
Number analyzed (sensor insertions) | 1528
percentage of successful insertion
  First 3 procedures: number analyzed (sensor insertions) | 102
  First 3 procedures | 100
  >3 procedures done: number analyzed (sensor insertions) | 1426
  >3 procedures done | 99.8
  Overall | 99.8

8. Secondary Outcome: Success Rate of Removal Procedures: Overall and by HCP Experience
Description: Success rate was measured for the first 3 removals for each inserting HCP, the remaining removals, as well as overall removals.
Time Frame: up to 27 months
Population: The number analyzed in the first 2 rows are the subsets of the overall removals based on HCP experience.
Measure: Number; unit: percentage of successful removals
Units Other Than Participants: sensor removals
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
Number analyzed (sensor removals) | 1517
percentage of successful removals
  First 3 procedures: number analyzed (Participants) | 102
  First 3 procedures | 96.1
  >3 procedures done: number analyzed (sensor removals) | 1415
  >3 procedures done | 98.7
  Overall | 98.4

9. Secondary Outcome: Rate of Insertion Procedures With Serious Adverse Events
Time Frame: up to 27 months
Measure: Count of Units; unit: insertions
Units Other Than Participants: insertions
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
Number analyzed (insertions) | 1528
insertions | 1

10. Secondary Outcome: Rate of Removal Procedures With Serious Adverse Events
Time Frame: up to 27 months
Measure: Count of Units; unit: removals
Units Other Than Participants: removals
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
Number analyzed (removals) | 1517
removals | 0

11. Secondary Outcome: HCP Feedback Questionnaire Regarding Insertion
Description: The questions were on a scale of 1-5, with 1 indicating Strongly Agree and 5 indicating Strongly Disagree.
Time Frame: up to 27 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
score on a scale
  The insertion procedure was easy | 1.1 (0.4)
  The labeling for use of the blunt dissector and the insertion tool are easy to understand | 1.1 (0.4)
  The blunt dissector and insertion tool are easy to use | 1.1 (0.3)
  The training was reflective of what I encountered during the insertion procedure | 1.2 (0.5)

12. Secondary Outcome: HCP Feedback Questionnaire Regarding Removal
Description: The questions were on a scale of 1-5, with 1 indicating Strongly Agree and 5 indicating Strongly Disagree.
Time Frame: up to 27 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
score on a scale
  The removal procedure was easy | 1.5 (0.8)
  The instructions and labeling for the removal were easy to understand | 1.2 (0.5)
  The clamp was easy to use to remove the sensor | 1.5 (0.7)
  The training was reflective of what I encountered during the removal procedure | 1.4 (0.7)

13. Secondary Outcome: Residual Dexamethasone Level in Explanted Sensors
Description: The residual dexamethasone (DXA) content in Sensors was analyzed after removal.
Time Frame: up to 27 months
Measure: Mean (Standard Deviation); unit: percentage of residual DXA
Arm/Group | Continuous Glucose Monitoring Device
Number analyzed (Participants) | 273
percentage of residual DXA | 82.5 (5.2)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from enrollment until study participation completion (approximately 27 months). Adverse events were followed until resolution, AE had stabilized, or the study had been completed. All AEs were adjudicated by CEC members.
Description: The reported adverse events are reported by number of sensor insertion cycles.
Arm/Group | Continuous Glucose Monitoring Device
All-Cause Mortality (participants affected / at risk) | 0/273
Serious Adverse Events (participants affected / at risk) | 21/273
Other Adverse Events (participants affected / at risk) | 115/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Monitoring Device (N=273)
Depression requiring hospitalization (Psychiatric disorders) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 1 (1)
Fracture of tibia and fibula (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoglycemic episode (Endocrine disorders) | 5 (8)
Hypoglycemia w/acute metabolic encephalopathy (Endocrine disorders) | 1 (1)
Acute stroke with ataxia (Nervous system disorders) | 1 (1)
Diabetic Ketoacidosis (Endocrine disorders) | 4 (4)
Cellulitis, bilateral lower extremity (Skin and subcutaneous tissue disorders) | 1 (1)
Foot infection, left (Musculoskeletal and connective tissue disorders) | 1 (1)
Congestive heart failure exacerbation (Cardiac disorders) | 2 (2)
Subdural hemorrhage (Nervous system disorders) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1)
COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Acute on chronic systolic heart failure (Cardiac disorders) | 1 (1)
Hyperglycemic hyperosmolar nonketotic (Endocrine disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Infection, Sensor insertion site (Infections and infestations) | 1 (1)
Myxedema crisis (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Monitoring Device (N=273)
Abdominal pain, gastritis, constipation (Gastrointestinal disorders) | 1 (1)
Abdominal pain, post-operative (Nervous system disorders) | 1 (1)
Abscess, right buttock (Skin and subcutaneous tissue disorders) | 1 (1)
Adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Immune system disorders) | 1 (1)
Ankle sprain, left (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Axillary swelling, post insertion (Immune system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bicep tear, right (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral Corneal Abrasions (Eye disorders) | 1 (1)
Bilateral Thumb Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bleeding, insertion site (Skin and subcutaneous tissue disorders) | 3 (3)
Blepharitis, bilateral (Eye disorders) | 1 (1)
Blister, foot (Skin and subcutaneous tissue disorders) | 1 (1)
Blistering, sensor insertion site (Skin and subcutaneous tissue disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bruise, sensor insertion site (Immune system disorders) | 2 (2)
Bump on left wrist (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis, bilateral shoulders (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis, left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis, left olecranon (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis, shoulder, right (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis, worsening (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataracts, left eye (Eye disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis, insertion site post removal (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis, insulin pump site, left hip (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis, left elbow (Skin and subcutaneous tissue disorders) | 1 (1)
Cholelithiasis (Gastrointestinal disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Cold sweat (Nervous system disorders) | 1 (1)
Concussion (Nervous system disorders) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
Contusion, left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Contusion, left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 17 (19)
Cracked tooth requiring extraction (General disorders) | 1 (1)
Deep venous thrombosis (Immune system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis, adhesive patch location (Skin and subcutaneous tissue disorders) | 2 (4)
Dermatitis, due to dermabond (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetic neuropathy, worsening (Nervous system disorders) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1)
Diaphoresis (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Dizziness (Vascular disorders) | 2 (2)
Dry eye syndrome (Eye disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea, worsening (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Reproductive system and breast disorders) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 1 (1)
Edema, bilateral lower extremities (Vascular disorders) | 1 (1)
Elbow fracture, left (Musculoskeletal and connective tissue disorders) | 1 (1)
Elbow fracture, right (Musculoskeletal and connective tissue disorders) | 1 (1)
Erythema, adhesive patch location (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema, sensor insertion site (Skin and subcutaneous tissue disorders) | 1 (1)
Fall with nasal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatty liver (Gastrointestinal disorders) | 1 (1)
Fecal impaction (Gastrointestinal disorders) | 1 (1)
Frozen shoulder, right (Musculoskeletal and connective tissue disorders) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 2 (2)
Head inury (General disorders) | 1 (1)
Headache/Migraine (Nervous system disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Heel pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatitis A exposure (Gastrointestinal disorders) | 1 (1)
Herpes Zoster infection (Skin and subcutaneous tissue disorders) | 1 (1)
Herpes zoster, eyelid (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidemia, worsening (Endocrine disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertension, worsening (Vascular disorders) | 2 (2)
Hypoglycemia (Endocrine disorders) | 3 (7)
Hypothyroidism, worsening (Endocrine disorders) | 1 (1)
Impetigo (Skin and subcutaneous tissue disorders) | 1 (1)
Infection, left eye (Eye disorders) | 1 (1)
Infection, sensor insertion site (Skin and subcutaneous tissue disorders) | 4 (4)
Influenza (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Insomnia (Nervous system disorders) | 1 (1)
Ischemia (Vascular disorders) | 1 (1)
Laceration, chin (Skin and subcutaneous tissue disorders) | 1 (1)
Laceration, upper lip (General disorders) | 1 (1)
Laryngeal papilloma, bilateral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lateral Epicondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Left jaw nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Left Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 2 (2)
Lipoma, paraspinal (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower extremity edema, bilateral (Vascular disorders) | 1 (1)
Lower respiratory tract infection, viral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lumbago exacerbation (Musculoskeletal and connective tissue disorders) | 1 (1)
Macular edema, left (Eye disorders) | 1 (1)
Marginal ulcer (Gastrointestinal disorders) | 1 (1)
Meniscal tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Menorragia (Reproductive system and breast disorders) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Mild Depression (Psychiatric disorders) | 1 (1)
Muscle strain, lower back (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle strain, ribcage (Metabolism and nutrition disorders) | 1 (1)
Nasal fracture (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Nausea and diarrhea, due to Covid-19 (Gastrointestinal disorders) | 1 (1)
Obstructive sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Onchomycosis (Skin and subcutaneous tissue disorders) | 1 (1)
Onychocryptosis, bilateral (Skin and subcutaneous tissue disorders) | 1 (1)
Oral surgery (Surgical and medical procedures) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Osteoarthritis, right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis, spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Endocrine disorders) | 1 (1)
Otitis Media (Ear and labyrinth disorders) | 1 (1)
Pain, sensor location (Nervous system disorders) | 5 (5)
Pain, sensor insertion site (Nervous system disorders) | 3 (3)
Pain, sensor removal site (Nervous system disorders) | 3 (3)
Panic attack (Psychiatric disorders) | 1 (1)
Paroxysmal Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Patellar fracture, closed, right (Musculoskeletal and connective tissue disorders) | 1 (1)
Pedal edema, bilateral (Cardiac disorders) | 1 (1)
Penile discharge (Reproductive system and breast disorders) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Phlebitis, superficial, bilateral (Vascular disorders) | 1 (1)
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Possible rabies exposure (Immune system disorders) | 1 (1)
Proliferative Retinopathy requiring Rx (Eye disorders) | 1 (1)
Prolonged wound healing (Skin and subcutaneous tissue disorders) | 1 (1)
Prolonged wound healing, removal site (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritis, adhesive patch location (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis, insertion site (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriatric arthritis, worsening (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Radiculopathy, cervical (Nervous system disorders) | 1 (1)
Rash, axilla and trunk (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, insertion site (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, lower extremities (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory infection due to Covid-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Restless arm syndrome (Nervous system disorders) | 1 (1)
Retinal tear, right (Eye disorders) | 1 (1)
Retinopathy, proliferative, bilateral (Eye disorders) | 1 (1)
RLS, worsened (Nervous system disorders) | 1 (1)
Scar, removal site (Skin and subcutaneous tissue disorders) | 3 (3)
Scarring, insertion site (Skin and subcutaneous tissue disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Sensor broke during removal (Product Issues) | 2 (2)
Sensor Location Site - Redness (Skin and subcutaneous tissue disorders) | 1 (1)
Sensory deficit, left heel (Nervous system disorders) | 1 (1)
Seroma, post surgical (Immune system disorders) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin atrophy, sensor site (Skin and subcutaneous tissue disorders) | 4 (4)
Skin depigmentation and atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discoloration, sensor site (Skin and subcutaneous tissue disorders) | 5 (6)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation, adhesive patch location (Skin and subcutaneous tissue disorders) | 4 (4)
Skin irritation, sensor insertion site (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation, sensor removal site (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep disturbance (Nervous system disorders) | 1 (1)
Sprain, left ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Sprain, neck and back (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Strep throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Swelling, incision site (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling, insertion site (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling, right foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Symptomatic Hyperglycemia (Endocrine disorders) | 1 (1)
Tendonitis, finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Tennis elbow, left (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombophlebitis, superficial, right arm (Immune system disorders) | 1 (1)
Thumb fracture, right (Musculoskeletal and connective tissue disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Toe fractures, right (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth fracture (General disorders) | 1 (1)
Tooth infection (General disorders) | 3 (4)
Torn meniscus, left (Musculoskeletal and connective tissue disorders) | 1 (1)
Torn meniscus, right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Transaminitis (Gastrointestinal disorders) | 1 (1)
Tremor, right hand (Nervous system disorders) | 1 (1)
Unable to remove sensor on first attempt (Surgical and medical procedures) | 20 (22)
Unstable angina (Cardiac disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Urinary tract infection (Renal and urinary disorders) | 4 (5)
Varicose veins, bilateral (Vascular disorders) | 1 (1)
Vasovagal episode (Nervous system disorders) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1)
Vibrating sensation at removal site (Immune system disorders) | 1 (1)
Vitamin D deficiency (Endocrine disorders) | 2 (2)
Vitreous detachment, right eye (Eye disorders) | 1 (1)
Vitreous syneresis, left eye (Eye disorders) | 1 (1)
Weakness, right arm (Nervous system disorders) | 1 (1)
Wrist fracture, left (Musculoskeletal and connective tissue disorders) | 2 (2)
Yeast infection, vaginal (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03908125/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT03908125/SAP_001.pdf